CLINICAL TRIAL: NCT02815319
Title: A Single Centre Randomised Study Comparing Standard of Care Schedules of Dexamethasone in Patients Incorrectly Taking Dexamethasone Premedication Prior to Docetaxel Chemotherapy (REaCT-dexamethasone)
Brief Title: Schedules of Dexamethasone in Patients Incorrectly Taking Dexamethasone Premedication (REaCT-dexamethasone)
Acronym: REaCT-dex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT 16-02
Record Dates: First submitted 2016-05-02; First posted 2016-06-28 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cancer
Keywords: Dexamethasone; Chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): Physician's treatment recommendation for dexamethasone premedication
  Interventions: Drug: Dexamethasone
- 8mg PO dexamethasone (Active Comparator): 8mg PO dexamethasone premedication
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Steroid prophylaxis
  Other Names: Decadron

SUMMARY:
Docetaxel chemotherapy is commonly used in patients with breast cancer. With the widespread use of steroid premedication, the incidence of fluid retention and skin toxicity side effects has been minimal. Premedication with dexamethasone (8mg twice daily) is recommended starting the day before chemotherapy and continuing for three days. Patients may forget to take all or part of their premedication prior to docetaxel administration, and additional doses of steroids are frequently give in place of the forgotten oral dose. The processes around treating patients who have incorrectly taken their medication are cumbersome leading to significant delays in patients receiving their chemotherapy while the chemotherapy nurse tries to contact the patients treating physician for guidance on the dose and route of dexamethasone they want administered. Most importantly with the current standard of care procedure, by the time the chemotherapy nurse, pharmacist and medical oncologist have spoken and made a treatment plan, the patient has been waiting for on average of an additional 1-2 hours before actually starting their chemotherapy.

DETAILED DESCRIPTION:
This study will randomize cancer patients to a standard dose of dexamethasone 8mg orally or to contact the physician to see what dose they recommend. The current trial proposal could therefore reduce the time for which patients are waiting to receive their chemotherapy, improving time patients need to spend in the hospital and significantly improving practice not just in Ottawa but globally.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving docetaxel chemotherapy for cancer
* Have incorrectly taken some or all of their dexamethasone premedication
* ≥19 years of age

Exclusion Criteria:

* Contraindication to dexamethasone
* Unable to give informed consent
* Already included in the study during a prior cycle

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
8mg PO stat is associated with significant reduction in time to commence docetaxel chemotherapy | 1 year
  To demonstrate that use of a standard replacement dose of dexamethasone (8mg PO stat) is associated with a significant reduction in the time for patients to commence their docetaxel chemotherapy.

SECONDARY OUTCOMES:
Hypersensitivity rate | 2 years
  Rates of hypersensitivity reactions to docetaxel
Fluid retention | 2 years
  Number of participants with fluid retention
Hospital cost | 2 years
  The hospital cost for each patient encounter will be estimated using a standardized case-costing methodology that was developed by the Ontario Case Costing Initiatives. This case-costing method is based on the Canadian Institute for Health Information Management Information Systems guidelines. The case-costing system links financial, clinical and patient activity information stored within information systems of the data warehouse to define "intermediate products" (e.g., nursing time, medications, laboratory tests). Direct and indirect hospital costs for each intermediate product used during an encounter are then summed for each patient.
Skin toxicity | 2 years
  Number of participants with skin toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Tina Hsu, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hsu T, Fergusson D, Stober C, Daigle K, Moledina N, Vandermeer L, Pond G, Hilton J, Hutton B, Clemons M; REaCT investigators. A randomized clinical trial comparing physician-directed or fixed-dose steroid replacement strategies for incomplete dexamethasone dosing prior to docetaxel chemotherapy. Support Care Cancer. 2021 Jun;29(6):3113-3120. doi: 10.1007/s00520-020-05791-5. Epub 2020 Oct 15. PMID 33057999